CLINICAL TRIAL: NCT01210131
Title: Individualized Hypoxia-guided Radiotherapy Combined With Standard Cisplatin-etoposide in Stage I-III SCLC
Brief Title: Hypoxia-guided Radiotherapy With Cisplatin-etoposide in Stage I-III : Small Cell Lung Cancer(SCLC)
Acronym: HX4 in SCLC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX4 in small cell lung cancer; 2010-023033-30 (EudraCT Number)
Record Dates: First submitted 2010-09-21; First posted 2010-09-28 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-01

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Toxicity; Progression; Survival; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma; Disease Progression | interventions — 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]HX4 (Experimental)
  Interventions: Drug: [18F]HX4

INTERVENTIONS:
Drug: [18F]HX4 — Intravenous injection

SUMMARY:
Since radiation dose escalation to a large volume of tumour inevitably will induce higher toxicity than is currently the case, efforts must be made to limit the volume of tissue irradiated. Moreover, the irradiation of larger tumour volumes leads to a lower achievable tumour dose when keeping the normal tissue doses constant. Central is thus the question whether it would be possible to limit the volume of tumour to be boosted by selectively escalating the radiation dose to specific disease sites which are theoretically more prone to relapse.

DETAILED DESCRIPTION:
Hypoxic imaging with PET scans seems attractive for this purpose as hypoxia is associated with resistance for radiotherapy and approximately 70 % of SCLC are severely hypoxic at diagnosis[2].

We hypothesize that it might be possible to use a selective boost in these patients to tumor areas which are still hypoxic at the end of the standard chemo-radiotherapy to a dose of 45 Gy in 30 fractions in 3 weeks.

This way all SCLC (small cell lung cancer) patients can receive a safe, but higher dose of radiotherapy to the whole tumor volume, while the most resistant areas receive the highest possible dose.

This is a hypothesis generating trial designed to deliver at least the current standard treatment to malignant tissue while defining patient selection criteria for future study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage I-III small cell lung cancer. WHO performance status 0-2
* Absolute neutrophil count at least 1800/µl and platelets at least 100000/µl and hemoglobin at least 6.2 mmol/l.
* Adequate renal function: calculated creatinine clearance at least 40 ml/min
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution (in case of liver metastases ≤ 5 x ULN for the institution)
* No previous platinum chemotherapy or topo-isomerase-inhibitors for SCLC.
* Lung function: FEV1 at least 30 % and DLCO at least 30 % of the age predicted value
* No history of prior chest radiotherapy
* Life expectancy more than 6 months
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant or breast feeding and willing to take adequate contraceptive measures during the study
* Ability to give and having given written informed consent before patient registration
* No mixed pathology, e.g. non-small cell plus small cell cancer
* No recent (< 3 months) severe cardiac disease (NYHA class >1) (congestive heart failure, infarction)
* No uncontrolled infectious disease
* No other active malignancy
* No major surgery (excluding diagnostic procedures like e.g. mediastinoscopy) in previous 4 weeks
* No treatment with investigational drugs in 4 weeks prior to or during this study

Exclusion Criteria:

* The opposite of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative local progression 18 months post-treatment as evaluated in a chest FDG-PET-CT scan | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival at two years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands